CLINICAL TRIAL: NCT00981747
Title: A Clinical Treatment Trial Targeting Vascular Reactivity in Idiopathic Pulmonary Fibrosis
Brief Title: Targeting Vascular Reactivity in Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding was withdrawn.
Sponsor: Alicia Gerke (Other)
Collaborators: Pulmonary Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Alicia Gerke, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200906736
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — Sildenafil Citrate; Losartan; Sugars

STUDY DESIGN:
Intervention Model Description: Participants will receive sildenafil for three months then losartan for three months, then sildenafil and losartan for three months and then placebo for three months in a random order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All study participants (Experimental): Study participants are patients that have been diagnosed with idiopathic pulmonary fibrosis (IPF).
  Interventions: Drug: Sildenafil; Drug: Losartan; Drug: Sildenafil and Losartan; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 20mg three times per day for 3 months followed by a one month washout prior to next intervention.
  Other Names: Viagra; Revatio
Drug: Losartan — Losartan 25mg two times a day for 3 months followed by a one month washout prior to next intervention.
  Other Names: Cozaar: losartan
Drug: Sildenafil and Losartan — Sildenafil 20mg three times per day and Losartan 25mg two times per day followed by a one month washout prior to next intervention.
  Other Names: Viagra, Revatio: sildenafil; Cozaar: losartan
Drug: Placebo Oral Tablet — Placebo pill three times per day for 3 months followed by a one month washout prior to next intervention.
  Other Names: Placebo pill (sugar)

SUMMARY:
The purpose of this study is to determine whether combination therapy with sildenafil and losartan can improve function and exercise tolerance in patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
It is currently suspected that the fibrosis in IPF is based upon an abnormal reparative process in the lung. Normally, an insult to the endothelium or epithelium of the lung would trigger an inflammatory process to help repair the site of injury; epithelial and endothelial cells then replicate and repair the tissue damage. In pulmonary fibrosis, alterations in this cascade change the balance of the inflammatory products and reduce the regulatory response which can produce continued inflammation. Fibrosis results from continued deposition of collagen by proliferating fibroblasts and lack of collagen breakdown.

In addition to fibrosis and microvascular destruction, pulmonary hypertension in IPF patients is a significant contributor to morbidity and mortality. The prevalence ranges from 32-85%, suggesting that pulmonary vascular disease is one of several processes that contribute to severity of disease.

We propose use of two therapeutic agents that affect the balance of vasoconstriction and vasodilation to improve basal tone of the vasculature. First, we propose the use of a phosphodiesterase inhibitor. Sildenafil (Viagra, Revatio) is an orally administered vasodilator that prolongs the effect of nitric oxide by inhibiting phosphodiesterase type 5 (PDE-5) which is responsible for degradation of cGMP. Increased cGMP concentration results in pulmonary vasculature relaxation and consequent vasodilation. Second, the use of an angiotensin receptor blocker (ARB) acts to diminish the direct vasoconstrictor effect of angiotensin and endothelin-1 in the vessels. In treatment of systemic hypertension, ARBs have been shown to be associated with a decrease in the amount of circulating endothelin-1 and increase in basal nitric oxide release. They have also been shown to rapidly inhibit the generation of reactive oxygen species by inflammatory cells. We test these interventions in a randomized cross-over trial in IPF patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99
* Have not taken any of the study medications in the past 6 weeks
* Diagnosed with idiopathic pulmonary fibrosis

Exclusion Criteria:

* FVC<50%, DLco <30% or FEV1/FVC ratio <65%
* Greater amount of emphysema than fibrotic change on chest CT scan
* Acute myocardial infarction within the past 6 months
* Nitrate use
* Contraindications, hypersensitivity, or allergic reaction to any study medication
* Presence of aortic stenosis
* Life-threatening arrhythmia within 1 month of evaluation
* Diabetes requiring insulin therapy
* Second-degree or third-degree atrioventricular block on electrocardiogram
* Echocardiographic evidence of severe pulmonary hypertension (>50mmHg) • Severe terminal illness (survival predicted to be less than 1 year)
* Severe congestive heart failure
* Renal impairment (creatinine >2.0 mg/dl)
* Moderate to severe hepatic impairment
* Concurrent treatment with immunosuppressive, cytotoxic, or investigational agents.
* Pregnant or Breastfeeding (Women of childbearing age must use effective form of birth control or abstinence during study participation)
* History of acute exacerbation of IPF
* Current enrollment in another investigational protocol
* Acute or chronic impairment other than dyspnea that limits the patient's ability to perform the six minute walk test
* Current drug or alcohol dependence
* Initiation of pulmonary rehabilitation within 30 days of enrollment. Subjects currently undergoing maintenance pulmonary rehabilitation at study entry will be asked to maintain their levels of rehabilitation for the duration of the trial
* Treatment of pulmonary hypertension with prostaglandins, endothelin-1 antagonists, or any other phosphodiesterase inhibitor within 30 days of enrollment
* Addition or discontinuation of calcium channel blockers, digitalis, diuretics or vasodilators within 30 days of enrollment. Dosage must be stable for 7 days prior to enrollment (except for diuretics)
* Listed for lung transplantation
* Due to drug interactions, all of the following agents will be prohibited: alpha-blockers, endothelin-1 antagonists, and CYP3A4 inhibitors
* Resting oxygen saturation of <92% with greater than 6 liters of supplemental oxygen

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia K Gerke, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Participants will be randomized to take one of the study medications (Sildenafil, Losartan, placebo oral tablet, and Sildenafil and Losartan) at a time. Participants will be randomized to take these medications for 3 months with a washout period of one month before starting the next medication. The order or medications taken is random in order to blind the investigator and participant
Period: Losartan
Arm/Group | All Study Participants
Started | 12
Started Losartan | 12
Completed Losartan | 10 (Only 9 were analyzed because only 9 completed all four interventions.)
Completed | 10 (Only 9 were analyzed because only 9 completed all four interventions.)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Period: Placebo Oral Tablet
Arm/Group | All Study Participants
Started | 10
Started Placebo Oral Tablet | 10
Completed Placebo Oral Tablet | 9
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Sildenafil
Arm/Group | All Study Participants
Started | 9
Started Sildenafil | 9
Completed Sildenafil | 9
Completed | 9
Not Completed | 0
Period: Sildenafil and Losartan
Arm/Group | All Study Participants
Started | 9
Started Sildenafil and Losartan | 9
Completed Sildenafil and Losartan | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects were randomized to complete all four arms in random order. There were nine participants analyzed in the study and all nine of those subjects participated in each arm. The numbers above do not include the 3 withdrawn subjects that did not complete the arms.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 63 [45 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Six Minute Walk Distance in Meters
Description: Change in 6MWD before and after treatment compared to placebo
Time Frame: At baseline and three months post each intervention.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Sildenafil: Sildenafil: Sildenafil 20mg three times per day for 3 months
- Losartan: Losartan: Losartan 25mg two times a day for 3 months
- Sildenafil and Losartan: Sildenafil and Losartan: Sildenafil 20mg three times per day and Losartan 25mg two times per day.
- Placebo: Placebo pill: Placebo pill three times per day for 3 months
Arm/Group | Sildenafil | Losartan | Sildenafil and Losartan | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
meters | 10.5 (23.1) | 15.8 (24.0) | -11.1 (12.0) | 12.1 (23.8)

2. Secondary Outcome: Change in Forced Vital Capacity (FVC)
Description: Change in FVC before and after treatment compared to placebo. FVC is a measure of lung size.
Time Frame: At baseline and three months post each intervention.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Sildenafil | Losartan | Sildenafil and Losartan | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
liters | -0.04 (.13) | -0.06 (0.13) | 0.002 (0.14) | -0.02 (0.14)

3. Secondary Outcome: Change in Shortness of Breath (SOB) Score
Description: Change in symptoms of SOB as determined by St. Georges Respiratory Questionnaire score. This score ranges from 0 to 100 with a higher score indicating more problems breathing.
Time Frame: At baseline and three months post each intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sildenafil | Losartan | Sildenafil and Losartan | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale | 2.1 (10.3) | 1.5 (5.7) | 3.3 (11.6) | -3.0 (9.8)

ADVERSE EVENTS:
Arm/Group | Sildenafil | Losartan | Sildenafil and Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/12 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/12 | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 7/9 | 9/12 | 7/9 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=9) | Losartan (N=12) | Sildenafil and Losartan (N=9) | Placebo (N=10)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Idiopathic Pulmonary Fibrosis Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Evaluated and documented idiopathic pulmonary fibrosis exacerbation confirmed by medical records.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=9) | Losartan (N=12) | Sildenafil and Losartan (N=9) | Placebo (N=10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2) — Increase or worsening of cough
Flushing (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Low blood pressure
Respiratory infection/viral illness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Outpatient treatment (no hospitalization)
Sinusitis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Not requiring hospitalization.

LIMITATIONS AND CAVEATS:
The trial was terminated early due to funding issues. Therefore, power to find a difference is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No